CLINICAL TRIAL: NCT04925011
Title: An Open-label, One-center Study Investigating the Efficacy and Safety of Roxadustat (FG-4592) for Treatment of Anemia in Pediatric Patients With Chronic Kidney Disease
Brief Title: Investigating the Efficacy and Safety of Roxadustat (FG-4592) for Treatment of Anemia in Pediatric Patients With CKD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mao Jianhua (Other)
Responsible Party: Sponsor-Investigator, Mao Jianhua, Chief Physician, The Children's Hospital of Zhejiang University School of Medicine
Organization: The Children's Hospital of Zhejiang University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Roxadustat for pediatric CKD
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Anemia Associated With Chronic Kidney Disease
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Roxadustat (Other): Starting doses of 20, 50, 70 or 100 mg/30,70,90,or 120mg based on weight and dialysis or not.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Starting doses of 20, 50, 70 or 100 mg/30,70,90,or 120mg based on weight and dialysis or not.

SUMMARY:
This open-labeled, one-center study is designed to evaluate the efficacy and safety of roxadustat in ESA-naïve and ESA-treated pediatric patients with CKD Stages 3, 4, and 5 who are receiving dialysis or not. The study will enroll patients between the ages of 2 to <18 years. Approximately 30 patients will be enrolled.

DETAILED DESCRIPTION:
This study is to evaluate the use of roxadustat for renal anemia in pediatric patients with CKD

ELIGIBILITY:
Inclusion Criteria:

1. Estimated glomerular filtration rate (Bedside Schwartz formula) of < 60 ml/min/1.73 m2 (stage 3, 4 and 5 CKD) for dialysis or non-dialysis patients.
2. For ESA-naïve patients, mean of two most recent central laboratory Hb values during the screening period obtained at least 2 days apart must be < 11.0 g/dL. For patients currently receiving stable ESA dosing who will discontinue ESA and convert to roxadustat during study, mean of two most recent central laboratory Hb values during the screening period obtained at least 2 days apart must be ≥ 9.0 g/dL and ≤ 12.5 g/dL
3. Ferritin >50 ng/mL and transferrin saturation >10%

Exclusion Criteria:

1. Uncontrolled hypertension as judged by the principal investigator prior to screening.
2. Known hematologic disease related anemia (including PRCA)
3. Known malignancy within the past 5 years before screening.
4. History of severe anaphylaxis or known allergic to ingredient of roxadusta.
5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3x upper limit of normal (ULN) and total bilirubin (Tbili) ≤2x ULN(obtained from screening visit).
6. Serum folate and vitamin B12 > LLN and cannot be corrected (obtained from screening visit).
7. Any RBC transfusion during the past 4 weeks before screening.
8. Weight<10kg
9. Any prior exposure to roxadustat or any other HIF-PH inhibitor.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with mean Hb ≥ 11.0 g/dL | weeks 16-24
  After the use of roxadustat, the proportion of patients with mean Hb ≥ 11.0 g/dL

SECONDARY OUTCOMES:
Mean change in Hb | weeks 16-24

CONTACTS AND LOCATIONS:
Overall Officials: jianhua Map, MD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No